CLINICAL TRIAL: NCT00996489
Title: Post-approval of Coaptite® in the Treatment of Female Urinary Incontinence
Brief Title: This is a Post Approval Study of Coaptite® in the Treatment of Female Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1005185
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-01

CONDITIONS: Female Stress Urinary Incontinence Due to Intrinsic Sphincter Deficiency

ARMS (1):
- Coaptite (Experimental)
  Interventions: Device: Coaptite®

INTERVENTIONS:
Device: Coaptite® — Calcium hydroxylapatite particles suspended in an aqueous based gel carrier

SUMMARY:
This is a post approval study of Coaptite® in the treatment of female urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Has female stress urinary incontinence that is due to intrinsic sphincter deficiency
* Has a baseline pad weight of greater than or equal to 50 grams
* Has viable mucosal lining at likely site of injection (bladder neck)
* Is at least 18 years of age
* Understands and accepts the obligation and is logistically able to present for all scheduled study visits
* Signs written informed consent

Exclusion Criteria:

* Has had a previous treatment for urinary incontinence with a urethral bulking agent other than Coaptite® or collagen
* Has detrusor instability
* Has bladder neuropathy
* Has nocturnal enuresis (bed wetting)
* Has Grade II or III prolapsed bladder
* Has overflow or functional incontinence
* Has significant history of urinary tract infections without resolution
* Has current or acute conditions of cystitis or urethritis
* Has history of significant pelvic irradiation
* Is pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2008-01-08 (Actual); Primary Completion 2015-10-26 (Actual); Study Completion 2015-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Wetumpka, Alabama
  - Surprise, Arizona
  - Encinitas, California
  - Los Angeles, California
  - Oceanside, California
  - Orange, California
  - Templeton, California
  - Celebration, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Berwyn, Illinois
  - Evanston, Illinois
  - Overland Park, Kansas
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Rochester, New York
  - Akron, Ohio
  - Houston, Texas
  - Temple, Texas
  - Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 sites in the United States.
Pre-assignment Details: A total of 459 participants were screened, enrolled and treated in the study. Of these, 298 participants completed the 36-month study.
Groups:
- Coaptite: Participants received first coaptite injection of calcium hydroxylapatite particles suspended in an aqueous based gel carrier, at baseline visit (Month 0) within 60 days of pad weight confirmation and the dosage was decided by the physician which was required to bulk the urethra to achieve the clinically desired level of incontinence correction. If an additional injection was determined to be clinically necessary, based on investigator's clinical judgement, participants received additional coaptite injections during 36 months.
Period: Overall Study
Arm/Group | Coaptite
Started | 459
Completed | 298
Not Completed | 161
Not completed — Device failure | 45
Not completed — Discontinued | 116

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all participants enrolled who were exposed to the study device at least once.
Arm/Group | Coaptite
Number analyzed (Participants) | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 459
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American | 1
  Asian | 9
  Black | 8
  Caucasian | 406
  Hispanic | 33
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 459

OUTCOME MEASURES:

1. Primary Outcome: Incontinence Status as Assessed by Stamey Grade Score
Description: The Stamey grade classifies the severity stress incontinence and was calculated from the 4-day voiding diary using the four possible grades from 0-3. Grade 0: controlled urination, Grade 1: accidents with vigorous activity, for example, lifting weights, coughing, and sneezing, Grade 2: accidents with minimal activity, for example, walking and standing up, and Grade 3: accidents regardless of activity or position and that cannot be attributed to a specific activity. Higher the Stamey grade, the most severe leakage level was estimated. An average of 4 days for the final grade was recorded and rounded up, if necessary (for example, 2.5 was equal to Grade 3).
Time Frame: Baseline and Months 6, 12, 18, 24, 30, and 36
Population: The full analysis set (FAS) consisted of SES participants who had a baseline and at least one post-baseline observed or imputed primary effectiveness value. Participants who were evaluable for this measure at given time period for the arm were included in the category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coaptite
Number analyzed (Participants) | 458
score on a scale
  Baseline | 2.5 (0.7)
  Month 6: number analyzed (Participants) | 408
  Month 6 | 1.6 (1.1)
  Month 12: number analyzed (Participants) | 391
  Month 12 | 1.5 (1.2)
  Month 18: number analyzed (Participants) | 361
  Month 18 | 1.6 (1.2)
  Month 24: number analyzed (Participants) | 350
  Month 24 | 1.5 (1.2)
  Month 30: number analyzed (Participants) | 328
  Month 30 | 1.5 (1.2)
  Month 36: number analyzed (Participants) | 329
  Month 36 | 1.5 (1.2)

2. Primary Outcome: Number of Participants With One Point Improvement in Stamey Grade Scores up to Month 12
Description: as for outcome 1
Time Frame: Baseline up to Month 12
Population: The FAS consisted of SES participants who had a baseline and at least one post-baseline observed or imputed primary effectiveness value. The FAS, where 6 and 12 months follow up data for the participants was available.
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 382
participants | 171

3. Primary Outcome: Number of Participants Who Had at Least One Point Improvement in Stamey Grade Scores Compared to Baseline
Description: as for outcome 1
Time Frame: Months 6, 12, 18, 24, 30, and 36
Population: The FAS consisted of SES participants who had a baseline and at least one post-baseline observed or imputed primary effectiveness value. Participants who were evaluable for this measure at given time period for the arm were included in the category.
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 458
participants
  Month 6: number analyzed (Participants) | 408
  Month 6 | 229
  Month 12: number analyzed (Participants) | 391
  Month 12 | 234
  Month 18: number analyzed (Participants) | 361
  Month 18 | 208
  Month 24: number analyzed (Participants) | 350
  Month 24 | 221
  Month 30: number analyzed (Participants) | 328
  Month 30 | 200
  Month 36: number analyzed (Participants) | 329
  Month 36 | 199

4. Primary Outcome: Number of Participants With Change From Baseline in Stamey Grade Scores Over Time
Description: as for outcome 1
Time Frame: Baseline up to Months 6 and 12
Population: The FAS consisted of SES participants who had a baseline and at least one post-baseline observed or imputed primary effectiveness value.
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 458
participants
  Month 6 | 408
  Month 12 | 391

5. Primary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to Month 36
Population: The SES was the subset of all participants enrolled who were exposed to the study device at least once.
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 459
participants | 313

6. Secondary Outcome: Number of Participants Who Received Each of the Six Coaptite Injections
Description: Coaptite injection were given to any participant during the 36 months of evaluation.
Time Frame: Baseline up to Month 36
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 458
participants
  Received First Injection | 458
  Received Second Injection | 262
  Received Third Injection | 90
  Received Fourth Injection | 26
  Received Fifth Injection | 7
  Received Sixth Injection | 1

7. Secondary Outcome: Time to Coaptite Retreatment
Description: Time to additional coaptite treatment or any other alternative treatment for stress urinary incontinence was recorded to assess the durability of effect.
Time Frame: Baseline up to Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Coaptite
Number analyzed (Participants) | 458
days
  Injection 1 to 2: number analyzed (Participants) | 262
  Injection 1 to 2 | 150.1 (189.6)
  Injection 2 to 3: number analyzed (Participants) | 90
  Injection 2 to 3 | 212 (215.3)
  Injection 3 to 4: number analyzed (Participants) | 26
  Injection 3 to 4 | 227.1 (222.1)
  Injection 4 to 5: number analyzed (Participants) | 7
  Injection 4 to 5 | 164 (74.0)
  Injection 5 to 6: number analyzed (Participants) | 1
  Injection 5 to 6 | 105 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

8. Secondary Outcome: Number of Participants With Alternative Treatments for Incontinence
Description: Number of participants with alternative treatment such as kegel exercises, sling, sling/cystocele repair, surgery, permanent abdominal tube, intravesical botox, sling/graft, sling removal, estradiol vaginal cream, bladder neck suspension, tension free vaginal tape, biofeedback, polydimethylsiloxane injections, solifenacin orally, bladder specific control physical therapy, for stress urinary incontinence were assessed.
Time Frame: Baseline up to Month 6 and Months 6 to 12, 12 to 18, 18 to 24, 24 to 30, 30 to 36
Population: The SES was the subset of all participants enrolled who were exposed to the study device at least once.
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 459
participants
  Kegel Exercises: Month 0-6 | 1
  Kegel Exercises: Month 6-12 | 1
  Kegel Exercises: Month 12-18 | 0
  Kegel Exercises: Month 18-24 | 0
  Kegel Exercises: Month 24-30 | 0
  Kegel Exercises: Month 30-36 | 0
  Sling: Month 0-6 | 5
  Sling: Month 6-12 | 2
  Sling: Month 12-18 | 4
  Sling: Month 18-24 | 8
  Sling: Month 24-30 | 5
  Sling: Month 30-36 | 0
  Sling/Cystocele Repair: Month 0-6 | 1
  Sling/Cystocele Repair: Month 6-12 | 3
  Sling/Cystocele Repair: Month 12-18 | 0
  Sling/Cystocele Repair: Month 18-24 | 1
  Sling/Cystocele Repair: Month 24-30 | 1
  Sling/Cystocele Repair: Month 30-36 | 0
  Surgery: Month 0-6 | 0
  Surgery : Month 6-12 | 1
  Surgery: Month 12-18 | 0
  Surgery: Month 18-24 | 0
  Surgery: Month 24-30 | 0
  Surgery: Month 30-36 | 0
  Permanent Abdominal Tube: Month 0-6 | 0
  Permanent Abdominal Tube: Month 6-12 | 0
  Permanent Abdominal Tube: Month 12-18 | 0
  Permanent Abdominal Tube: Month 18-24 | 0
  Permanent Abdominal Tube: Month 24-30 | 0
  Permanent Abdominal Tube: Month 30-36 | 1
  Intravesical Botox: Month 0-6 | 0
  Intravesical Botox: Month 6-12 | 1
  Intravesical Botox: Month 12-18 | 1
  Intravesical Botox: Month 18-24 | 1
  Intravesical Botox: Month 24-30 | 2
  Intravesical Botox: Month 30-36 | 1
  Sling/Graft, Sling Removal: Month 0-6 | 0
  Sling/Graft, Sling Removal: Month 6-12 | 0
  Sling/Graft, Sling Removal: Month 12-18 | 0
  Sling/Graft, Sling Removal: Month 18-24 | 1
  Sling/Graft, Sling Removal: Month 24-30 | 0
  Sling/Graft, Sling Removal: Month 30-36 | 0
  Estradiol Vaginal Cream: Month 0-6 | 0
  Estradiol Vaginal Cream: Month 6-12 | 0
  Estradiol Vaginal Cream: Month 12-18 | 0
  Estradiol Vaginal Cream: Month 18-24 | 1
  Estradiol Vaginal Cream: Month 24-30 | 0
  Estradiol Vaginal Cream: Month 30-36 | 0
  Bladder Neck Suspension: Month 0-6 | 1
  Bladder Neck Suspension: Month 6-12 | 1
  Bladder Neck Suspension: Month 12-18 | 1
  Bladder Neck Suspension: Month 18-24 | 0
  Bladder Neck Suspension: Month 24-30 | 0
  Bladder Neck Suspension: Month 30-36 | 0
  Tension Free Vaginal Tape: Month 0-6 | 0
  Tension Free Vaginal Tape: Month 6-12 | 1
  Tension Free Vaginal Tape: Month 12-18 | 0
  Tension Free Vaginal Tape: Month 18-24 | 0
  Tension Free Vaginal Tape: Month 24-30 | 0
  Tension Free Vaginal Tape: Month 30-36 | 0
  Biofeedback: Month 0-6 | 1
  Biofeedback: Month 6-12 | 0
  Biofeedback: Month 12-18 | 0
  Biofeedback: Month 18-24 | 0
  Biofeedback: Month 24-30 | 0
  Biofeedback: Month 30-36 | 0
  Polydimethylsiloxane Injections: Month 0-6 | 0
  Polydimethylsiloxane Injections: Month 6-12 | 1
  Polydimethylsiloxane Injections: Month 12-18 | 0
  Polydimethylsiloxane Injections: Month 18-24 | 1
  Polydimethylsiloxane Injections: Month 24-30 | 0
  Polydimethylsiloxane Injections: Month 30-36 | 0
  Solifenacin orally: Month 0-6 | 0
  Solifenacin orally: Month 6-12 | 0
  Solifenacin orally: Month 12-18 | 0
  Solifenacin orally: Month 18-24 | 0
  Solifenacin orally: Month 24-30 | 0
  Solifenacin orally: Month 30-36 | 1
  Bladder SpecificControlPhysical TherapyX6:0-6 | 0
  BladderSpecificControlPhysicalTherapyX6:Month6-12 | 0
  BladderSpecificControlPhysicalTherapyX6:Month12-18 | 0
  BladderSpecificControlPhysicalTherapyX6:Month18-24 | 0
  BladderSpecificControlPhysicalTherapyX6:Month24-30 | 1
  BladderSpecificControlPhysicalTherapyX6:Month | 0

9. Secondary Outcome: Number of Participants With Urge Incontinence Medication (UIM) Status
Description: The use of urge incontinence medications was collected pre-treatment and post-treatment.
Time Frame: Baseline up to Month 36
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Coaptite
Number analyzed (Participants) | 427
participants | 52

10. Secondary Outcome: Incontinence Quality of Life (iQoL) Scores
Description: The iQoL measured the effect of urinary incontinence on QoL. It was divided into 3 subscales: 1 (avoidance and limiting behaviour); 2 (psychosocial impact), and 3 (social embarrassment). The iQOL was comprised of 22 items, each with the response scale from 1 (extremely) to 5 (not at all). A mean score for each subscale was calculated (averaging the scores for the items in each subscale) as well as a total score for all 22 items (sum of all subscale scores). The scores were then transformed to a scale score ranging from 0 to 100 points, where higher scores indicated less impact of incontinence on QoL.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, and 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaptite
Number analyzed (Participants) | 458
units on a scale
  Baseline: number analyzed (Participants) | 455
  Baseline | 39.5 (21.9)
  Month 6: number analyzed (Participants) | 411
  Month 6 | 69.6 (24.5)
  Month 12: number analyzed (Participants) | 398
  Month 12 | 70.3 (24.5)
  Month 18: number analyzed (Participants) | 371
  Month 18 | 70.4 (24.4)
  Month 24: number analyzed (Participants) | 357
  Month 24 | 71.2 (24.3)
  Month 30: number analyzed (Participants) | 334
  Month 30 | 73.5 (24.3)
  Month 36: number analyzed (Participants) | 330
  Month 36 | 72.7 (24.4)

11. Secondary Outcome: Volume of Coaptite Injected Per Treatment
Time Frame: Baseline, Baseline to Month 6 and Months 6 to 12, 12 to 18, 18 to 24, 24 to 30, 30 to 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Coaptite
Number analyzed (Participants) | 458
milliliter (mL)
  Baseline | 1.8 (0.7)
  Baseline to Month 6: number analyzed (Participants) | 264
  Baseline to Month 6 | 1.8 (0.8)
  Month 6 to 12: number analyzed (Participants) | 41
  Month 6 to 12 | 1.5 (0.6)
  Month 12 to 18: number analyzed (Participants) | 36
  Month 12 to 18 | 2.0 (0.7)
  Month 18 to 24: number analyzed (Participants) | 17
  Month 18 to 24 | 1.7 (0.8)
  Month 24 to 30: number analyzed (Participants) | 14
  Month 24 to 30 | 1.7 (0.8)
  Month 30 to 36: number analyzed (Participants) | 14
  Month 30 to 36 | 1.6 (1.3)

12. Secondary Outcome: Mean Number of Sites Injected by Coaptite
Time Frame: Baseline, Baseline to Month 6 and Months 6 to 12, 12 to 18, 18 to 24, 24 to 30, 30 to 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: number of sites
Arm/Group | Coaptite
Number analyzed (Participants) | 458
number of sites
  Baseline | 2.4 (0.9)
  Baseline to Month 6: number analyzed (Participants) | 264
  Baseline to Month 6 | 2.4 (0.9)
  Month 6 to 12: number analyzed (Participants) | 41
  Month 6 to 12 | 2.5 (0.9)
  Month 12 to 18: number analyzed (Participants) | 36
  Month 12 to 18 | 2.6 (1.0)
  Month 18 to 24: number analyzed (Participants) | 17
  Month 18 to 24 | 2.5 (1.0)
  Month 24 to 30: number analyzed (Participants) | 14
  Month 24 to 30 | 2.9 (1.8)
  Month 30 to 36: number analyzed (Participants) | 14
  Month 30 to 36 | 2.1 (0.3)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 36
Description: While the CRF was not designed to capture Serious Adverse Events (SAEs), following review of the safety data, Merz reported serious medical device reports (MDRs) to the FDA for 163 subjects and as a result, a subset of adverse events (AEs) originally classified as Other AEs were re-classified as SAEs. In some cases, the same adverse event term could correspond to either a serious or non-serious adverse event depending on the presence or absence of associated serious medical device report.
Arm/Group | Coaptite
All-Cause Mortality (participants affected / at risk) | 10/459
Serious Adverse Events (participants affected / at risk) | 163/459
Other Adverse Events (participants affected / at risk) | 246/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coaptite (N=459)
Urinary tract infection (Infections and infestations) | 114
Fungal infection (Infections and infestations) | 5
Cystitis (Infections and infestations) | 4
Vulvovaginal mycotic infection (Infections and infestations) | 2
Urinary retention (Renal and urinary disorders) | 63
Urge incontinence (Renal and urinary disorders) | 27
Micturition urgency (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 3
Nocturia (Renal and urinary disorders) | 2
Urethritis noninfective (Renal and urinary disorders) | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1
Cystocele (Reproductive system and breast disorders) | 2
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coaptite (N=459)
Urinary tract infection (Infections and infestations) | 136
Micturition urgency (Renal and urinary disorders) | 29
Urge incontinence (Renal and urinary disorders) | 109
Urinary retention (Renal and urinary disorders) | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.